CLINICAL TRIAL: NCT00226109
Title: Effect of Spironolactone Treatment on Heart- and Skeletal Muscle in Chronic Alcoholics
Brief Title: Clinical Trial Studying the Effects of Spironolactone on Heart and Skeletal Muscle Function in Chronic Alcoholics
Acronym: SPICA
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Problems recruting patients
Sponsor: University of Aarhus (Other)
Responsible Party: Peter Holland-Fischer, Department of Medicine V, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AFDV01; 01
Record Dates: First submitted 2005-09-23; First posted 2005-09-26 (Estimated); Last update posted 2010-10-20 (Estimated); Status verified 2010-10

CONDITIONS: Cardiomyopathy, Alcoholic; Alcoholism
Keywords: Alcoholism; cardiomyopathy; skeletal muscle; spironolactone; Na,K-pumps; Magnesium
MeSH Terms: conditions — Cardiomyopathy, Alcoholic; Alcoholism; Cardiomyopathies | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Active Comparator)
  Interventions: Drug: spironolactone

INTERVENTIONS:
Drug: spironolactone — 100 mg once daily. Can be reduced to 50 mg a day still maintaining the doubled-blinded status
  Other Names: Spirix; Spiron

SUMMARY:
Chronic alcoholics suffer from weak skeletal and cardiac muscle. The investigators have discovered a beneficial effect of spironolactone-treatment in that regard. Therefore, a double blind placebo controlled study is conducted, to examine the effects of spironolactone on cardiac and skeletal muscle-function in chronic alcoholics.

DETAILED DESCRIPTION:
Our department has done research into skeletal muscle function in patients with liver cirrhosis. Post-hoc analyses of one of these studies suggested that treatment with spironolactone had a positive effect on muscle strength and endurance. This effect was probably caused by an increase in concentration of Na, K-pumps (sodium-potassium pumps) enabling the muscle cell perform better.

To verify this finding we have designed a double-blinded, placebo-controlled, randomized clinical trial with skeletal muscle strength, -endurance, Na, K-pump content, cardiac systolic, and diastolic function as primary endpoints. Spironolactone is tested against placebo in 40 participants included among our admitted and out-clinic patients. Muscle function-tests, muscle biopsy and trans-thoracic echocardiography is performed before and after 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Alcoholism, male gender

Exclusion Criteria:

* Spironolactone treatment
* Tense ascites
* Hepatic encephalopathy
* Dementia
* Cancer
* Severe psychiatric disease
* Untreated thyroid disease
* Maltreated diabetes
* Spironolactone contraindications
* Kidney failure

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-04; Primary Completion 2011-08 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Muscle strength | 0 and 12 weeks
Muscle endurance | At 0 and 12 weeks
Content of Na,K-pump in skeletal muscle | 0 and 12 weeks
Content of sodium and potassium in skeletal muscle | 0 and 12 weeks
Steptest result | 0 and 12 weeks
Diastolic heart function | 0 and 12 weeks
Systolic heart function | 0 and 12 weeks

SECONDARY OUTCOMES:
Muscle mass | 0 and 12 weeks
QTc interval | 0 and 12 weeks
Magnesium retention | 0, 6, and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Vilstrup, Proffessor, Principal Investigator — Univeristy of Aarhus; Peter Holland-Fischer, MD, Study Director — University of Aarhus
Locations (1):
- Department of Medicine V (gastroenterology and hepatology), Aarhus, Denmark